CLINICAL TRIAL: NCT05932355
Title: Assessment of the Effect of Plasmid Inhibitors and Antimicrobial Drugs as Combined Strategy Against Clinical Multi-drug Resistant Hypervirulent Klebsiella Pneumoniae
Brief Title: Synergistic Effect of Plasmid Inhibitors and Antimicrobial Drugs Against Clinical MDR-hvKP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Elnokrashy Mohamed, Principal Investigator, Assiut University
Other Study IDs: Plasmid inhibitors in MDR-hvKP
Record Dates: First submitted 2023-05-15; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Synergy Between Plasmid Inhibitors and Combined Antibiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fifty Endotracheal aspirates will be collected aseptically from VAP patients admitted to chest ICU in Assiut University Hospital with immediate transport to Microbiology and Immunology department laboratories, Faculty of Medicine, Assiut University. Samples will be stored at -20 for further DNA extraction.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Screening for MDR-hvKP causing VAP in patients admitted to chest ICU in Assiut University Hospital.
2. In vitro evaluation of the synergistic activity of combined meropenem/levofloxacin with and without kasugamycin against clinical MDR-hvKP isolates by checkerboard and time killing assay.
3. In vivo evaluation of the synergistic activity of combined meropenem/levofloxacin with and without kasugamycin using MDR-hvKP septic rat model.

DETAILED DESCRIPTION:
New "hypervirulent" Klebsiella-pneumoniae (hvKp) strain has emerged as a clinically-significant-pathogen in both healthy and immunocompromised individuals . HvKp, at its discovery, was rarely resistant to antimicrobial-agents , however, nowadays, antibiotic-resistant hvKP isolates are being reported .

Plasmids are important vectors that bacteria use to transfer resistance and virulence determinants. Typically, genetic elements conferring resistance and virulence were encoded by different plasmids . Most recently, clinicians have been faced, the confluence of resistance and virulence-determinants on the same or coexisting-plasmids with the evolution of multidrug-resistant (MDR) and hypervirulent Klebsiella pneumoniae hvKP .

One approach to combat MDR infections is to combine antimicrobial drugs during a treatment-regimen . Fluoroquinolone plus carbapenems is one of-the most useful-combination used in cases which suffer from MDR to most available monotherapies . Another-approach is Plasmid curing, using plasmid inhibitors, which is the method of removing plasmids from the bacterial populations while leaving the population intact leading to reversal of the plasmid-mediated antibiotic resistance .

Kasugamycin, an-aminoglycoside; is a compound exhibiting significant-antiplasmid activity-up-to-complete suppression of plasmid-replication . Kasugamycin was found to block plasmid replication by inhibiting-expression of plasmid replication initiation-protein, RepE, and to reduce plasmid-levels by 90% . Accordingly, we hypothesize that, using dual-antibiotics supplemented with plasmid inhibitor will be efficient in inhibiting MDR-hvKP, both in vitro and in vivo.

This is the first-study to evaluate the effect of addition of plasmid inhibitor on improving the efficacy of antibiotics and improve their synergistic activity. The results of this study will open the door for-using plasmid-inhibitor-compounds on restoring the usefulness of many conventional-antibiotics to which-resistance has emerged.

ELIGIBILITY:
Inclusion Criteria:

VAP patients (patients under mechanical ventilation for more than 48 h with new or progressive infiltrate on chest X-ray and have at least two of the following criteria:

1. Fever (>38 oC) with no other recognized cause
2. WBCs < 4000/mm3 or >12000/mm3
3. New onset of purulent sputum.
4. Increase in respiratory secretion or increased need for suctioning.
5. New-onset or worsening cough, or dyspnea, or tachypnea worsening gas exchange.

Exclusion Criteria:

Patients with chest diseases other than VAP .

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Fifty VAP patients with no other chest diseases will be included in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Synergistic effect of plasmid inhibitors and antimicrobial drugs against MDR-hvKP invitro. | 24hours
  Assessment of synergy invitro by :
  Checkerboard assay : Fractional inhibitory concentrations index (FICI) will be calculated as:
  FICI = FIC A (MIC for antibiotic A in combination) / (MIC antibiotic A) + FIC B (MIC antibiotic B in combination) / (MIC antibiotic B). (It is a ratio)
  Synergy is defined as FICI ≤0.5, no interaction is defined as FICI > 0.5 and ≤ 4, and antagonism is defined as FICI >4 .
  .

CONTACTS AND LOCATIONS:
Overall Officials: Sherine Aly, Professor, Study Director — Department of Microbiology and Immunology; Wegdan Mohamad, Assistant Professor, Study Director — Department of Microbiology and Immunology

REFERENCES:
- [Background] Prokesch BC, TeKippe M, Kim J, Raj P, TeKippe EM, Greenberg DE. Primary osteomyelitis caused by hypervirulent Klebsiella pneumoniae. Lancet Infect Dis. 2016 Sep;16(9):e190-e195. doi: 10.1016/S1473-3099(16)30021-4. Epub 2016 Jul 9. PMID 27402393
- [Background] Zhang Y, Zhao C, Wang Q, Wang X, Chen H, Li H, Zhang F, Li S, Wang R, Wang H. High Prevalence of Hypervirulent Klebsiella pneumoniae Infection in China: Geographic Distribution, Clinical Characteristics, and Antimicrobial Resistance. Antimicrob Agents Chemother. 2016 Sep 23;60(10):6115-20. doi: 10.1128/AAC.01127-16. Print 2016 Oct. PMID 27480857
- [Background] Zhan L, Wang S, Guo Y, Jin Y, Duan J, Hao Z, Lv J, Qi X, Hu L, Chen L, Kreiswirth BN, Zhang R, Pan J, Wang L, Yu F. Outbreak by Hypermucoviscous Klebsiella pneumoniae ST11 Isolates with Carbapenem Resistance in a Tertiary Hospital in China. Front Cell Infect Microbiol. 2017 May 16;7:182. doi: 10.3389/fcimb.2017.00182. eCollection 2017. PMID 28560183
- [Background] Feng Y, Lu Y, Yao Z, Zong Z. Carbapenem-Resistant Hypervirulent Klebsiella pneumoniae of Sequence Type 36. Antimicrob Agents Chemother. 2018 Jun 26;62(7):e02644-17. doi: 10.1128/AAC.02644-17. Print 2018 Jul. PMID 29712659
- [Background] Worthington RJ, Melander C. Combination approaches to combat multidrug-resistant bacteria. Trends Biotechnol. 2013 Mar;31(3):177-84. doi: 10.1016/j.tibtech.2012.12.006. Epub 2013 Jan 18. PMID 23333434
- [Background] Drago L, De Vecchi E, Nicola L, Colombo A, Guerra A, Gismondo MR. Activity of levofloxacin and ciprofloxacin in combination with cefepime, ceftazidime, imipenem, piperacillin-tazobactam and amikacin against different Pseudomonas aeruginosa phenotypes and Acinetobacter spp. Chemotherapy. 2004 Oct;50(4):202-10. doi: 10.1159/000081033. Epub 2004 Sep 23. PMID 15452399
- [Background] Vrancianu CO, Popa LI, Bleotu C, Chifiriuc MC. Targeting Plasmids to Limit Acquisition and Transmission of Antimicrobial Resistance. Front Microbiol. 2020 May 6;11:761. doi: 10.3389/fmicb.2020.00761. eCollection 2020. PMID 32435238
- [Background] Zulauf KE, Kirby JE. Discovery of small-molecule inhibitors of multidrug-resistance plasmid maintenance using a high-throughput screening approach. Proc Natl Acad Sci U S A. 2020 Nov 24;117(47):29839-29850. doi: 10.1073/pnas.2005948117. Epub 2020 Nov 9. PMID 33168749